CLINICAL TRIAL: NCT04284319
Title: Heart Transplantation Using Normothermic Regional Perfusion (NRP) Donation After Circulatory Death (DCD): A Pilot Study
Brief Title: Heart Transplantation Using Normothermic Regional Perfusion Donation After Circulatory Death
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-01664
Record Dates: First submitted 2020-01-24; First posted 2020-02-25 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Heart Transplantation; Normothermic Regional Perfusion; NRP; Donation After Circulatory Death; DCD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCD Heart Transplantation Using NRP (Experimental): Heart Transplantation Using Normothermic Regional Perfusion (NRP) Donation After Circulatory Death (DCD)
  Interventions: Procedure: DCD Heart Transplantation Using NRP

INTERVENTIONS:
Procedure: DCD Heart Transplantation Using NRP — Heart Transplantation Using Normothermic Regional Perfusion (NRP) Donation After Circulatory Death (DCD)

SUMMARY:
Normothermic regional perfusion (NRP) utilizes Extracorporeal Membrane Oxygenation (ECMO) or cardiopulmonary bypass to reperfuse the heart and other organs in situ after isolation and ligation of the cerebral vessels. In situ resuscitation of the heart has the added advantage of allowing full hemodynamic and echocardiographic assessment of the donor heart prior to final acceptance for transplantation without the imminent danger of ongoing warm ischemia.

DETAILED DESCRIPTION:
The current procedure of DCD organ donation and procurement follows a well-established course for lung, liver, kidney and pancreas transplantation in the United States. After consent has been obtained, the organs are allocated through UNOS. When all parties are present and ready, the donor is withdrawn from life support (i.e., discontinuation of mechanical ventilation and any vasoactive medications). The surgical teams are generally present on the premises but not at the donor's bedside. After circulatory arrest occurs, which is determined by the absence of pulse and organized rhythmic cardiac activity, death is declared by a physician not associated with the transplant teams. Subsequently a period of stand-off is observed (5 minutes for organs donated in New York) to ensure complete cessation of the circulation before organ procurement is commenced. If after withdrawal of life support the patient does not progress to circulatory death within the allotted time (variable among hospitals, but 180 minutes in this study), the procurement is abandoned and the patient is transferred out of the operating room and placed on palliative measures.

Given that DCD organ donation is already currently practiced in the US, the same standard approach defined by each state and locality can also be applied to DCD heart donation and will be followed for this protocol at NYULH. However, this protocol will utilize a normothermic regional perfusion (NRP) strategy that involves reestablishment of circulatory blood flow after the period of circulatory arrest has been established and the 5 minutes of standoff time has passed. The local Organ Procurement Organization (LiveOnNY) and NYULH Medical Leadership have reviewed and approved this approach to DCD heart donation. Specifically, normothermic regional perfusion involves the following steps:

1. Opening the chest through a standard sternotomy used for heart and lung procurement.
2. Ligation of the all the blood vessels that supply blood to the brain to ensure that blood flow to the brain is not reestablished once circulation is restarted as described below.
3. Standard cannulation of the aorta and the right atrium as is done for cardiac surgical procedures.
4. Initiation of cardiopulmonary bypass, which will re-establish the flow of blood to all organs of the body including the heart under normothermia. The initial step for ligation of the blood vessels to the head is necessary to ensure that blood flow to the brain does not occur.

Once blood flow to the heart is established, the heart will start beating. At 30 minute intervals, the donor will be separated from cardiopulmonary bypass and the heart will be assessed for functionality. If accepted standard DBD procurement will commence. The heart transplantation surgery on the potential recipient will only begin once the heart has been accepted as suitable.

If after assessment the heart is not suitable, cardiopulmonary bypass will be restarted. The donor heart will be reassessed at 30 minute intervals up to 180 minutes. If no significant acceptable recovery occurs and the heart is not deemed suitable for transplantation, then the study will be terminated, but the remaining organs can be recovered as standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient is ≥ 18 years old
2. Recipient, or their designated healthcare proxy, is able and willing to sign informed consent
3. Recipient meets standard listing criteria for heart transplantation at NYU Langone Health Transplant Institute

Exclusion Criteria:

1. Recipient is < 18 years old
2. Recipient, or their designated healthcare proxy, is unable to sign informed consent
3. Recipient is participating in another interventional trial
4. Recipient has a known history of HIV infection
5. Recipient has any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Successful NRP-DCD Heart transplants | One Year
  The primary outcome is the rate of successful NRP-DCD heart transplants.

SECONDARY OUTCOMES:
Number of living authorized representatives who authorize candidate's organs for donation and research | One Year
Number of candidates who are transferred to NYU Langone Health for donation after circulatory death (DCD) | One Year
Number of candidates who progress to death after withdrawal of care | One Year
Number of Donors whose hearts are deemed suitable for donation following normothermic regional perfusion (NRP) | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Nader Moazami, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No